CLINICAL TRIAL: NCT07240441
Title: Endo-ePIcardial Versus Endocardial Only Catheter Ablation for ISchemic Driven Ventricular Tachycardia (EPISODE VT) - Multicenter, Prospective, Randomized Trial
Brief Title: Endo-ePIcardial Versus Endocardial Only Catheter Ablation for ISchemic Driven Ventricular Tachycardia (EPISODE VT)
Acronym: EPISODE_VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MEDICOVER SP Z O.O. (Other)
Collaborators: National Institute of Cardiology, Warsaw, Poland (Other); Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPISODE VT; 2024/ABM/01/00005 (Other Grant/Funding Number: MEDICAL RESEARCH AGENCY (AGENCJA BADAŃ MEDYCZNYCH - PL))
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Ventricular Tachycardias; Myocardial Infarction (MI); Implantable Cardiac Defibrillator; Ablation
Keywords: ventricular tachycardia; myocardial infarction; epicardial access; pericardial sac puncture; ablation; implantable cardioverter defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocardial post MI VT ablation group (Active Comparator): Endocardial post MI VT radiofrequency ablation using contact force irrigated catheters, standard electrophysiological systems, electroanatomical mapping systems and RF generators.
  Interventions: Procedure: Endocardial VT ablation
- Endo-epicaridal post MI VT ablation group (Experimental): Endo-epicardial post-myocardial infarction VT radiofrequency ablation will be performed using contact force irrigated catheters, standard electrophysiological systems, electroanatomical mapping systems and RF generators. Access to the pericardial sac will be preceded by CO2 insufflation into its lumen.
  Interventions: Procedure: Endo-epicardial VT ablation

INTERVENTIONS:
Procedure: Endocardial VT ablation — Post-myocardial infarction VT radiofrequency ablation using a standard endocardial approach
  Arms: Endocardial post MI VT ablation group
Procedure: Endo-epicardial VT ablation — Post-myocardial infarction VT radiofrequency ablation using an endo-epicardial approach with pericardial sac puncture preceded by CO2 insufflation
  Arms: Endo-epicaridal post MI VT ablation group

SUMMARY:
The EPISODE VT trial is designed to compare efficacy and safety of two modalities for interventional treatment - endocardial ablation and endo-epicardial ablation in a population of patients with post myocardial infarction (ICD 10 - I25.2) ventricular tachycardias (ICD 10 - I47.2), who are protected by an implantable cardioverter-defibrilator (ICD) and meet study inclusion criteria.

DETAILED DESCRIPTION:
The EPISODE VT trial is designed to compare efficacy and safety of two modalities for interventional treatment - endocardial ablation and endo-epicardial ablation in a population of patients with post myocardial infarction (ICD 10 - I25.2) ventricular tachycardias (ICD 10 - I47.2), who are protected by an implantable cardioverter-defibrilator (ICD) and meet study inclusion criteria. Nowadays, most often ablation is performed using only endocardial approach. The rate of VT recurrences after such ablation may exceed 50%, which is largely due to the inability to remove all arrhythmogenic substrate. At the same time, in cases where all potentially arrhythmogenic substrate is removed, the immediate and long-term results are better, both in terms of recurrence and prognosis. Single reports on endo-epicardial ablation as the first-line therapy in patients with post-infarction VT indicate a higher efficacy of this approach compared to endocardial ablation. Similar conclusions emerge from meta-analyses. This is probably due to a more complete removal of the arrhythmogenic substrate located mainly in the epicardium or intramurally.

In the endo-epicardial group pericardial sac puncture will be performed after filling it with carbon dioxide, which creates a space for safe puncture.

Ablation procedures will be performed as standard. The electrophysiological systems and ablation electrodes used in the study will be standard devices that research centers are equipped with. Their use will be in accordance with the procedures of the center and the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Status after myocardial infarction (minimum 3 months before inclusion in the study).
* Documented post-infarction VT or VF.
* Implantable ICD (at least 2 weeks before ablation) or CRT-D (at least 2 months before ablation).
* A history of at least one from below:

  1. One or more high energy interventions.
  2. Three or more adequate antitachycardia pacing therapies, including one symptomatic.
  3. Three or more episodes of VT in 24 hours (interrupted by ATP or shock) - electrical storm.
  4. Sustained VT recorded on ECG with a cycle length longer than the ICD detection threshold.
* Age between 18 and 85 years.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Obesity with BMI > 40 kg/m2.
* Left ventricle ejection fraction < 20%.
* Pregnancy or breastfeeding.
* Renal failure (eGFR < 20 mL/min/1.73m2).
* Fresh ballot thrombus in the left ventricle.
* Suspicion of massive adhesions in the pericardium that may impede pericardial puncture.
* Ablation of the post-infarction VT in the left ventricle in medical history.
* Previous heart surgery.
* Acute conditions that prevent ablation (including active infection, overt hyperthyroidism and others listed below).
* Active neoplastic disease.
* Heart failure with NYHA IV.
* Life expectancy less than 12 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 2 years
  Death from any cause
Electrical storm (3 episodes of VT in 24 hours) | 2 years
Adequate ICD shock during 24 months of follow-up. | 2 years

CONTACTS AND LOCATIONS:
Locations (9):
- Poland (9):
  - Medicover Hospital, Warsaw, Masovian Voivodeship
  - Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - National Institute of Cardiology, Warsaw, Masovian Voivodeship
  - University Hospital No. 1 in Bydgoszcz, Bydgoszcz
  - University Clinical Center based in Gdańsk, Gdansk
  - Independent Public Health Care Facility University Hospital in Krakow, Krakow
  - University Clinical Hospital in Poznań, Poznan
  - University Clinical Hospital No. 2 PUM in Szczecin, Szczecin
  - Grochowski Hospital named after Dr. Rafał Masztak, MD, Warsaw

IPD SHARING:
Plan to Share IPD: No